CLINICAL TRIAL: NCT04492631
Title: A 4-Week Study to Evaluate the Safety of a Probiotic Water Containing Streptococcus Salivarius DB-B5 in Healthy Volunteer Subjects
Brief Title: Safety of an Oral Probiotic in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dose Biosystems Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: P1940120
Record Dates: First submitted 2020-07-17; First posted 2020-07-30 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Powdered probiotic with a carrier.
  Interventions: Dietary Supplement: Streptococcus salivarius DB-B5
- Placebo (Placebo Comparator): Carrier only.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Streptococcus salivarius DB-B5 — Sachets containing Streptococcus salivarius DB-B5 will be dissolved in water and consumed by the participants (n=30) once daily for 4 weeks. The participants will consume 10 billion colony forming units (CFU) per day.
  Arms: Probiotic
Other: Placebo — Sachets containing a placebo (probiotic carrier) will be dissolved in water and consumed by the participants (n=30) once daily for 4 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of an oral probiotic in healthy individuals.

DETAILED DESCRIPTION:
The oral cavity houses one of the most diverse microbiota in the human body. There are nearly 800 unique oral bacterial species identified with more species expected to be added with further sampling and identification. As with microbiota of other sites in the human body, a balanced oral microbiota is essential to maintaining the health of the human host. Streptococcus salivarius is a pioneer species that colonizes the human oral cavity from birth, and remains a predominant member of the commensal microbiota throughout life. This randomized, double-blind, placebo-controlled study is conducted to investigate the safety and tolerability of a Streptococcus salivarius DB-B5 strain.

ELIGIBILITY:
Inclusion Criteria:

1. Are adults, 18 to 65 years of age and in good general health and good oral health (no active or uncontrolled diseases or conditions);
2. Have a body mass index (BMI) range of 18.5 - 35 kg/m^2;
3. Have no known food allergies or intolerances;
4. Have normal or acceptable to the Investigator vital signs (blood pressure, heart rate, respiratory rate, temperature) at screening and Day -1 and normal laboratory values and physical exam findings at screening;
5. Agree not to make any major changes to their diet during the study;
6. Read and sign the Research Subject Information and Consent Form;
7. Are willing to use the assigned products according to instructions, attend scheduled appointments, and complete the study;
8. Are males and females who agree to use medically acceptable contraception (oral/implant/injectable/transdermal contraceptives, intrauterine device, condom with spermicide, diaphragm with spermicide, abstinence, partner's vasectomy, tubal ligation; abstinence or vasectomies are acceptable if the female subject agrees to implement two of the other acceptable methods of birth control if her lifestyle/partner changes) for the duration of the study and 30 days after study completion and attest to having used it for three months prior to screening, if of child-bearing potential;
9. If subject is a female of child-bearing potential, agrees to submit to a urine pregnancy test (UPT) at screening, Day -1 and at the end of study / early termination visit.

Exclusion Criteria:

1. Have self-reported history of active or chronic dental or medical disease;
2. Are prone to gas, bloating, or diarrhea;
3. Have received antibiotic treatment in the three months prior to Day 1 or are unwilling to refrain from antibiotic use during the study;
4. Used probiotic supplements or consumed probiotic rich foods such as yogurt or kefir within 30 days prior to Day 1 or are unwilling to refrain from the use of probiotic supplements or probiotic rich foods for the duration of the study, even if they are for non-oral health reasons (e.g., vaginal or gut health probiotics);
5. Are pregnant, planning to become pregnant during the study period, or are breastfeeding a child;
6. Self-reported current users of tobacco products, vaping products, cannabis, and/or nicotine replacement therapy (gums, lozenges, sprays, etc.);
7. Frequent users of alcohol, defined as consumption of 21 units or more of alcoholic beverage per week (21 units = 6 L of beer, 2.5 L of wine, or 500 mL of spirits);
8. Used over-the-counter (OTC) laxatives or any other medications, supplements, or products that, in the opinion of the Investigator, could influence the endpoints in this study within 30 days prior to Day 1 or are unwilling to refrain from the use of these products for the duration of the study;
9. Have chronic or acute illness such as heart disease, diabetes, cancer, autoimmune conditions, or history of human immunodeficiency virus (HIV) that, in the opinion of the Investigator, could impact the outcome of the study;
10. Have any other condition or situation that may increase the risk associated with study participation or may interfere with the study results, in the opinion of the Investigator;
11. Are unwilling or unable to provide informed consent and follow study procedures;
12. Have participated in any clinical study within the 30 days prior to Day 1;
13. Are clinical site personnel or relative or partner of clinical site personnel.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
Reports of adverse events | 4 weeks
  Reports of adverse events will be collected and compared between the probiotic and placebo groups.
Change in gastrointestinal symptoms measured using the Gastrointestinal Symptom Rating Scale (GSRS) | 4 weeks
  Gastrointestinal tolerability to the test products will be assessed using the Gastrointestinal Symptom Rating Scale (GSRS). The GSRS is composed of 15 items covering 5 dimensions: Reflux, Abdominal pain, Indigestion, Diarrhea and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
Occurrence of abnormal blood laboratory test results | 4 weeks
  Fasting blood samples will be collected at baseline and end-of-study visits to assess for changes in hematology parameters (complete blood count including differentials and platelets).
Occurrence of abnormal clinical chemistry parameters test results | 4 weeks
  Fasting blood samples will be collected at baseline and end-of-study visits to assess for changes in clinical chemistry parameters (basic metabolic panel, hepatic function panel).
Occurrence of abnormal urinalysis test results | 4 weeks
  Urine samples will be collected at baseline and end-of-study visits to assess for changes in standard urinalysis parameters (specific gravity, pH, ketones, glucose, blood, bilirubin, and leukocyte esterase).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Casser, M.D., Principal Investigator — TKL Research, Inc.
Locations (1):
- TKL Research, Inc., Fair Lawn, New Jersey, United States

REFERENCES:
- [Derived] Li X, Fields FR, Ho M, Marshall-Hudson A, Gross R, Casser ME, Naito M. Safety assessment of Streptococcus salivarius DB-B5 as a probiotic candidate for oral health. Food Chem Toxicol. 2021 Jul;153:112277. doi: 10.1016/j.fct.2021.112277. Epub 2021 May 15. PMID 34004226